CLINICAL TRIAL: NCT06576752
Title: Contemporary Post-Discharge Management in Heart Failure At Home
Brief Title: Management of Patients with Heart Failure At Home After Hospital Discharge
Acronym: STRONG@HOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Drammen sykehus (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Peder L. Myhre, MD, PhD, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 721190
Record Dates: First submitted 2024-08-13; First posted 2024-08-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: heart failure; digital health; remote monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home care (Experimental): Follow-up and management of HF medications at home visits after 1, 2, 3 and 6 weeks performed by telecommunication led by HF nurses in close communication with physician at the institution. Around week 2 a single visit to the primary care physician's office is required.
  Interventions: Other: Digital follow-up and uptitration of medications at home after hospital discharge for heart failure
- Hospital care (Active Comparator): Follow-up and management of HF medications provided by specialists at the participating institutions' outpatient clinics after 1, 2, 3 and 6 weeks. (Same as the high-intensity arm in STRONG-HF)
  Interventions: Other: Follow-up and uptitration of medications at the hospital outpatient-clinic after hospital discharge for heart failure

INTERVENTIONS:
Other: Digital follow-up and uptitration of medications at home after hospital discharge for heart failure — Both arms will treat the patients according to the STRONG-HF intensive care strategy, as recommended by current guidelines. That is up-titration to at least half of maximum tolerated doses of HF medications at discharge, followed by up-titration to maximum tolerated doses after 2 weeks. Safety visits will be performed after 1, 3 and 6 weeks.
  Other Names: Dignio (digital healthcare platform); Checkware (digital healthcare platform); Nimble (digital healthcare platform)
  Arms: Home care
Other: Follow-up and uptitration of medications at the hospital outpatient-clinic after hospital discharge for heart failure — Both arms will treat the patients according to the STRONG-HF intensive care strategy, as recommended by current guidelines. That is up-titration to at least half of maximum tolerated doses of HF medications at discharge, followed by up-titration to maximum tolerated doses after 2 weeks. Safety visits will be performed after 1, 3 and 6 weeks.
  Arms: Hospital care

SUMMARY:
This study aims to assess whether patients with acute heart failure (HF) can achieve the same level of HF-therapies by digital follow-up at home as compared to hospital visits according to the STRONG-HF strategy. Patients admitted to hospital with acute HF will be enrolled and randomized to either follow-up at the hospital out-patient clinic or digital follow-up at home.

DETAILED DESCRIPTION:
This study seeks to enhance the management of HF patients by demonstrating that follow-up and medication up-titration can be effectively carried out digitally at home, thereby relieving the burden on healthcare systems and patients. There exists a substantial knowledge gap in the implementation of life-saving HF drugs that have been shown to significantly reduce mortality in HF patients, by as much as 73%. Despite strong evidence from clinical trials and guidelines, the utilization of optimal HF therapy among patients remains low. The successful STRONG-HF trial demonstrated improved outcomes through early and rapid up-titration of HF medications and follow-up at specialized HF clinics after discharge, and this strategy is now strongly recommended in the updated European Society of Cardiology Heart Failure Guidelines from 2023. However, a major challenge was the need for patients to travel to the hospital for weekly visits, which posed significant barriers for many patients, especially in geographically dispersed regions due to travel distance, immobility, and logistical challenges. To address this gap, the STRONG@HOME trial aims to conduct visits and rapid up-titration of medications in the patient's home, a strategy not previously tested in a clinical trial and with direct clinical implications. The success of this approach has the potential to improve HF care globally and advance the field of implementation science in HF and other chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission within the 72 hours prior to screening for acute HF.
* NT-proBNP > 1,500 pg/mL measured during the hospitalization
* Systolic blood pressure ≥ 100 mmHg and of heart rate ≥ 60 bpm within 24 hours before randomization
* Serum potassium ≤ 5.0 mEq/L (mmol/L).
* ≤ ½ the optimal dose of ACEi/ARB/ARNi or beta-blocker or MRA.
* Written informed consent to participate in the study.

Exclusion Criteria:

1. Age below 18 or above 85 years.
2. Clearly documented intolerance to high doses of beta-blockers
3. Clearly documented intolerance to high doses of renin-angiotensin system (RAS) blockers (both ACEi and ARB).
4. Renal disease or estimated glomerular filtration rate (eGFR) below 30 mL/min/1.73m2 at screening or history of dialysis.
5. Prior (defined as less than 30 days from screening) or current enrollment in a HF intervention or participation in an investigational drug or device study within the 30 days prior to screening
6. Index event (admission for acute HF) triggered primarily by a completely reversable etiology so that it is unlikely the patient will be classified with chronic HF after discharge, such as Takotsubo syndrome (stress cardiomyopathy). In the setting of acute coronary syndrome or tachycardia, this should be managed before considering the presence of HF. This does not apply to patients with chronic HF prior to the index event.
7. Severe non-adherence to medications
8. Psychiatric or neurological disorder, cirrhosis, or active malignancy leading to a life expectancy less than 6 months.
9. History of heart transplant or on a transplant list, or using or planned to be implanted with a ventricular assist device.
10. Uncorrected thyroid disease, active myocarditis, or known amyloid or hypertrophic obstructive cardiomyopathy.
11. Inability to comply with all study requirements, due to major co-morbidities, social or financial issues, or a history of noncompliance with medical regimens, that might compromise the patients ability to understand and/or comply with the protocol instructions or follow-up procedures.
12. Low digital competency classified as inability to handle a smartphone or tablet.
13. Language barriers requiring the need for an external interpreter.
14. Pregnant or nursing (lactating) women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Guideline recommended medical treatment Score (0-9) | 90 days
  Patients are assigned a score for each of the four drug classes, and the sum of these is the total score. For beta-blockers and ACEi/ARBs, patients are assigned 0 (no treatment), 1 (<50% target daily dose), or 2 points (≥50% target daily dose) for each therapy. Any dose of ARNI instead of ACEi/ARB are assigned 3 points. Any dose of MRA and SGLT2i are assigned 2 points. Proportion of patients with ≥50% dose of ACEi/ARB/ARNI, MRA and beta blocker and treatment with SGLT2i
Treatment-emergent adverse events | 90 days
  Proportion of patients with eGFR of <30 mL/min/1.73 m2, systolic BP of <95 mm Hg, heart rate of <50 bpm, and serum potassium of >5.5 mmol/L.

SECONDARY OUTCOMES:
Achieved dose in each of the components of the primary endpoint (mg) | 90 days
  Renin-angiotensin-system blockers, mineralocorticoid receptor antagonists and beta blockers, and treatment with sodium-glucose cotransporter-2-inhibitors
Proportion of patients with baseline LVEF<40% with ≥50% dose of guideline recommended heart failure medications | 90 days
  Proportion of patients with ≥50% dose of renin-angiotensin-system blockers, mineralocorticoidreceptor antagonists and beta blockers, and treatment with sodium-glucose cotransporter-2-inhibitors in the subgroup with baseline left ventricular ejection fraction<40%
Change in quality of life by EQ-5D index | 90 days
  Measured by EuroQol Group (EQ-5D) index questionnaire (range 11111 to 55555, higher is worse)
Change in quality of life by EQ-5D VAS | 90 days
  Measured by EuroQol Group (EQ-5D) questionnaire (range 0 to 100, lower is worse)
Change in N-terminal pro-B-type natriuretic peptide (ng/L) | 90 days
  From baseline
Change in echocardiographic measures of left ventricular structure | 90 days
  Left ventricular end diastolic volume index (ml/m^2)
Change in body weight (kg) | 90 days
  From baseline
Self-care | 90 days
  European Heart Failure Self-care Behaviour [EHFScB] scale (range 9-45, higher is worse)
Patient satisfaction with digital follow-up | 90 days
  IT-HEART questionnaire (range 10-50, higher is worse)
Number of heart failure readmissions | 12 months and 24 months
  Admissions to the hospital for heart failure
Number of total readmissions | 12 months and 24 months
  All admissions to the hospital
Time out of hospital | 12 months and 24 months
  Days not admitted to a hospital after baseline
Number of deaths | 12 months and 24 months
  All-cause mortality
Cost | 90 days, 12 months, 24 months
  To evaluate the total cost of each follow up strategy by summarizing the cost of healthcare utilization, digital platform costs and travel costs
Change in HF-specific quality of life | 90 days
  Minnesota Living with HF questionnaire (range 0-105, higher is worse)
Change in echocardiographic measure of cardiac diastolic function | 90 days
  E/e' (ratio)
Change in echocardiographic measure of cardiac systolic function | 90 days
  Left ventricular ejection fraction (%)

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog, Akershus
  - Drammen Hospital, Vestre Viken HF, Drammen, Vestre Viken

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data

REFERENCES:
- [Background] Mebazaa A, Davison B, Chioncel O, Cohen-Solal A, Diaz R, Filippatos G, Metra M, Ponikowski P, Sliwa K, Voors AA, Edwards C, Novosadova M, Takagi K, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G. Safety, tolerability and efficacy of up-titration of guideline-directed medical therapies for acute heart failure (STRONG-HF): a multinational, open-label, randomised, trial. Lancet. 2022 Dec 3;400(10367):1938-1952. doi: 10.1016/S0140-6736(22)02076-1. Epub 2022 Nov 7. PMID 36356631